CLINICAL TRIAL: NCT01199458
Title: The Effect of Alfentanil on the Lower Esophageal Sphincter During Anesthesia Induction - a Study in Volunteers
Brief Title: The Effect of an Opioid on the Lower Esophageal Sphincter During Anesthesia Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT nr: 2010-020697-41
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2010-09

CONDITIONS: Lower Esophageal Sphincter
Keywords: Lower Esophageal Sphincter; Barrier pressure
MeSH Terms: interventions — Alfentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- opioid (Active Comparator): Preoxygenation for 5 min. Injection of opioid (alfentanil 20 mikrogr/kg iv) after 2 min:Injection of induction drug(propofol 2-2.5mg/kg) after anesthesia induction: Application of cricoid pressure for 15 sec.
  Interventions: Drug: alfentanil
- placebo (Placebo Comparator): Preoxygenation for 5 min. Injection of saline iv. after 2 min:Injection of induction drug(propofol 2-2.5mg/kg) after anesthesia induction: Application of cricoid pressure for 15 sec.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: alfentanil — 20 mikrogr/kg
  Other Names: alfentanil = rapifen
  Arms: opioid
Drug: saline — The amount of saline will be equal the amount (in ml) of the study-drug (alfentanil)in order to keep it blinded.
  Arms: placebo

SUMMARY:
This study evaluates the effects of adding an opioid (alfentanil) during anesthesia induction with respect to the barrierpressure in the esophagogastric junction.

The secondary aim was to investigate whether the effect of cricoid pressure influences the barrierpressure.

DETAILED DESCRIPTION:
During anesthesia induction and tracheal intubation one major concern is to avoid passive regurgitation of gastric content and aspiration.

The lower esophageal sphincter is a muscle located at the distal end of the esophagus. It plays an important role in creating a barrier between the stomach and the esophagus. The term "barrierpressure" is defined as the pressure difference between the lower esophageal sphincter pressure and the pressure in the stomach (intragastric pressure).

There are studies showing that opioids given iv/im, in the vein or in the muscle, may decrease the pressure in the lower esophageal sphincter and hereby increase the risk of aspiration.

Nevertheless,other studies shows that opioids are still frequently given to patients during anesthesia induction. This is done in order to prevent the cardiovascular response to (the painful) intubation which can often be seen as an equally high risk for the patient as the risk of aspiration.

In light of the above description, the investigators are planning a study in volunteers with the primary aim of investigating the effects of an opioid (alfentanil) on the pressures in the lower esophageal sphincter.

Another safety measure taken during anesthesia induction is the so called "cricoid pressure". This is based on the theory that passive regurgitation of gastric content may be prevented by occluding the esophagus by pressing on the cricoid cartilage. However, there are studies indicating that the application of cricoid pressure also may decrease the tonus of the lower esophageal sphincter.

The secondary aim of the study is to investigate the effect of cricoid pressure application on the pressure in the lower esophageal sphincter.

Measurements are being done using high-resolution solid-state manometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer 18-40 years old
* Informed,signed and dated consent

Exclusion Criteria:

* Pharyngoesophageal dysfunction
* Gastro/intestinal-,cardiovascular-,lung- or neurologic disease
* Ongoing medication
* Allergy to alfentanil, propofol, soya or peanuts
* Pregnancy or breast-feeding
* BMI>30
* Participation in other clinical trial -ongoing or during last 30 days.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Changes in barrierpressure (in mmHg) in the area of the lower esophageal sphincter. | 1 min after the application of the induction agent (propofol)
  Pressure variations in the lower esophageal sphincter will be measured continuously during the whole study. Registrations will be saved in the computer-software. Predetermined time points will be marked on the registrations for later evaluation.

SECONDARY OUTCOMES:
Changes in barrierpressure (in mmHg) in the area of the lower esophageal sphincter. | during cricoidpressure application (continues for 15 sec)
  Pressure variations in the lower esophageal sphincter will be measured continuously during the whole study. Registrations will be saved in the computer-software. Predetermined time points will be marked on the registrations for later evaluation.
Changes in barrierpressure (in mmHg) in the area of the lower esophageal sphincter. | 1min after the opioid/placebo injection
  Pressure variations in the lower esophageal sphincter will be measured continuously during the whole study. Registrations will be saved in the computer-software. Predetermined time points will be marked on the registrations for later evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wattwil, MD PhD, Principal Investigator — Department of Anesthesia and Intensive Care, Örebro University Hospital, Örebro,Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Original data can be available by contacting the principal investigator